CLINICAL TRIAL: NCT00387257
Title: A Double Blind, Placebo Controlled, Parallel Study to Evaluate Effects of Repeat Doses of Rilapladib on Platelet Aggregation in Healthy Male Volunteers
Brief Title: Effect Of Rilapladib (SB-659032) On Platelet Aggregation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: LP2108364
Record Dates: First submitted 2006-10-10; First posted 2006-10-12 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-04

CONDITIONS: Healthy Subjects; Atherosclerosis
Keywords: platelet aggregation; SB-659032; rilapladib
MeSH Terms: conditions — Atherosclerosis | interventions — rilapladib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Rilapladib (SB-659032)

SUMMARY:
The purpose of this study is to compare the effects of repeat doses of SB-659032 with placebo on platelet aggregation in subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with QTc < 450 msec as measured at screening.

Exclusion Criteria:

* History of asthma.
* Smokers.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2006-10; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Collagen EC50 values on Day 35 (or 21 days post last dose) as determine by optical aggregometry. | on Day 35 (or 21 days post last dose) as determine by optical aggregometry

SECONDARY OUTCOMES:
Collagen EC50 values on Day 1 and Day 14 as determined by optical aggregometry Plasma Lp-PLA2 activity Clinical safety data Concentrations of rilapladib and SB-664601. | on Day 1 and Day 14 as determined by optical aggregometry

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Randwick, New South Wales, Australia

REFERENCES:
- [Derived] Shaddinger BC, Xu Y, Roger JH, Macphee CH, Handel M, Baidoo CA, Magee M, Lepore JJ, Sprecher DL. Platelet aggregation unchanged by lipoprotein-associated phospholipase A(2) inhibition: results from an in vitro study and two randomized phase I trials. PLoS One. 2014 Jan 27;9(1):e83094. doi: 10.1371/journal.pone.0083094. eCollection 2014. PMID 24475026